CLINICAL TRIAL: NCT05207956
Title: App for Strengthening Services In Specialized Therapeutic Support
Acronym: ASSISTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 849995
Record Dates: First submitted 2021-11-24; First posted 2022-01-26 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Data collection; autism; Behavioral Health Technician (BHT); behavioral economics; implementation; implementation strategy; implementation science; Therapeutic Support Staff (TSS)
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: After consenting to participate in the trial, participants will be randomized in pairs to one of the two study arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Electronic Platform (Experimental): A basic electronic platform for data collection that contains additional features designed to increase motivation to collect data and ease of data collection.
  Interventions: Behavioral: Behavioral economics strategies; Other: Electronic platform
- Electronic Platform Not Enhanced (Active Comparator): A basic electronic platform for data collection.
  Interventions: Other: Electronic platform

INTERVENTIONS:
Behavioral: Behavioral economics strategies — Behavioral economics features designed to increase motivation to collect data and ease of data collection on the electronic platform.
  Arms: Enhanced Electronic Platform
Other: Electronic platform — Electronic platform to collect data

SUMMARY:
In partnership with a digital health software company, the University research team created two versions of a mobile application to help behavioral health technicians (BHT's) who work with students with autism collect data. The first version comprises a basic electronic platform for data collection. The second version has the same basic electronic platform for data collection, plus additional features designed to increase motivation to collect data and ease the burden of data collection.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be working as a paraprofessionals or behavioral health technicians
* Currently providing individual support to children with autism
* Currently providing services in Philadelphia preschools, schools, day cares, or homes.

Exclusion Criteria:

* n/a

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enhanced Electronic Platform | Electronic Platform Not Enhanced
Started | 14 | 13
Completed | 13 | 11
Not Completed | 1 | 2
Not completed — Lost to follow up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Electronic Platform | Electronic Platform Not Enhanced | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.5 (10.2) | 41.6 (14.6) | 38.6 (12.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 6 | 3 | 9
  Female | 7 | 10 | 17
  Non-binary/ third gender | 0 | 0 | 0
  Prefer not to disclose | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 13 | 12 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 6 | 12
  White | 5 | 7 | 12
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 14 | 13 | 27
Work experience, Years [Mean (Standard Deviation); unit: years] | 5.4 (4.5) | 7.4 (4.6) | 6.4 (4.55)

OUTCOME MEASURES:

1. Primary Outcome: The Difference in Data Collection Consistency Between Groups Across Three Weeks
Description: Consistency was the percentage of intervals in which aides entered data per session with children during each school day, across a three week period. These metrics were captured via web analytics in partnership with our digital health company.
Time Frame: Three-week trial period
Population: 27 were enrolled (14 treatment, 13 control) and data complete for 23
Measure: Mean (95% Confidence Interval); unit: percentage of intervals
Arm/Group | Enhanced Electronic Platform | Electronic Platform Not Enhanced
Number analyzed (Participants) | 13 | 11
percentage of intervals | .66 [.51 to .80] | .44 [.19 to .70]

2. Primary Outcome: The Difference in Data Collection Completion Between Groups Across Three Weeks
Description: as for outcome 1
Time Frame: Three-week trial period
Population: 27 were enrolled (14 treatment, 13 control) and data was complete for 23
Measure: Mean (95% Confidence Interval); unit: percentage of intervals
Arm/Group | Enhanced Electronic Platform | Electronic Platform Not Enhanced
Number analyzed (Participants) | 13 | 10
percentage of intervals | .81 [.67 to .96] | .98 [.96 to 1.00]

3. Primary Outcome: The Difference in Data Collection Timeliness Between Groups Across Three Weeks
Description: as for outcome 1
Time Frame: Three-week trial period
Population: 27 were enrolled (14 treatment, 13 control) and data was complete for 22
Measure: Mean (95% Confidence Interval); unit: percentage of intervals
Arm/Group | Enhanced Electronic Platform | Electronic Platform Not Enhanced
Number analyzed (Participants) | 12 | 10
percentage of intervals | 4.69 [1.76 to 7.62] | 71.87 [-9.32 to 153.05]

4. Secondary Outcome: Intentions for Implementors
Description: We adapted scales to measure mechanisms affecting data collection, including intentions, using social psychology methods (Armitage & Connor, 2001). The intentions measure had one item, which was rated from 1=strongly disagree to 7=strongly agree. Strongly agree meant stronger intentions to take data. Aides completed measures at baseline and post-trial (3 weeks). Data reported are changes over time.
Time Frame: Assessed at baseline and end of 3-week trial period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Electronic Platform | Electronic Platform Not Enhanced
Number analyzed (Participants) | 13 | 11
score on a scale | 5.31 (2.59) | 5.91 (2.07)

5. Secondary Outcome: System Usability Scale
Description: We used the System Usability Scale (SUS; Brooke, 1996) to measure aides' reactions to various statements regarding the app's usability with 10 items that use a 5-point scale from (1) strongly disagree to (5) strongly agree. The SUS has high internal consistent reliability (Cronbach's alpha = .91) and demonstrated sensitivity to change (Lewis, 2018). We adapted the original questionnaire to replace "system" with "app" across all items. The SUS is calculated as a proportion score out of 100, with higher scores indicating higher usability (≥85 = Excellent; ≥71 = Good; ≥51 = Okay (Bangor et al.).
Time Frame: Three-week trial period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Electronic Platform | Electronic Platform Not Enhanced
Number analyzed (Participants) | 13 | 11
score on a scale | 76.4 (15.2) | 67.7 (21.5)

6. Secondary Outcome: Attitudes for Implementors
Description: We adapted scales to measure mechanisms affecting data collection, including attitudes, using social psychology methods (Armitage & Connor, 2001). The attitudes measure had one item, which was rated from 1=good to 7=bad (meaning that taking data would be bad). Attitudes had 2 items. These items were averaged to create the scale score which could range from 1 to 7 for each measure. Aides completed measures at baseline and post-trial (3 weeks). Data reported are changes over time.
Time Frame: Assessed at baseline and end of 3-week trial period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Electronic Platform | Electronic Platform Not Enhanced
Number analyzed (Participants) | 13 | 11
score on a scale | 6.54 (1.03) | 6.68 (0.73)

7. Secondary Outcome: Perceived Norms for Implementors
Description: We adapted scales to measure mechanisms affecting data collection, including perceived norms, using social psychology methods (Armitage & Connor, 2001). The perceived norms measure had one item, which was rated from 1=strongly disagree to 7=strongly agree. Strongly agree meant stronger influence of norms on taking data. Aides completed measures at baseline and post-trial (3 weeks). Data reported are changes over time.
Time Frame: Assessed at baseline and end of 3-week trial period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Electronic Platform | Electronic Platform Not Enhanced
Number analyzed (Participants) | 13 | 11
score on a scale | 5.62 (2.14) | 6.18 (1.83)

8. Secondary Outcome: Descriptive Norms for Implementors
Description: We adapted scales to measure mechanisms affecting data collection, including descriptive norms, using social psychology methods (Armitage & Connor, 2001). The perceived norms measure had one item, which was rated from 1=strongly disagree to 7=strongly agree. Strongly agree meant stronger influence of norms on taking data. Aides completed measures at baseline and post-trial (3 weeks). Data reported are changes over time.
Time Frame: Assessed at baseline and end of 3-week trial period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Electronic Platform | Electronic Platform Not Enhanced
Number analyzed (Participants) | 13 | 11
score on a scale | 6.08 (1.60) | 6.27 (1.27)

9. Secondary Outcome: Self-Efficacy for Implementors
Description: We adapted scales to measure mechanisms affecting data collection, including self-efficacy, using social psychology methods (Armitage & Connor, 2001). The self-efficacy measure had one item, which was rated from 1=strongly disagree to 7=strongly agree. Strongly agree meant stronger self-efficacy about taking data. Self-Efficacy had 2 items. These items were averaged to create the scale score which could range from 1 to 7 for each measure. Aides completed measures at baseline and post-trial (3 weeks). Data reported are changes over time.
Time Frame: Assessed at baseline and end of 3-week trial period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Electronic Platform | Electronic Platform Not Enhanced
Number analyzed (Participants) | 13 | 11
score on a scale | 5.5 (1.72) | 4.91 (2.50)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the three week trial period for every participant.
Description: The University of Pennsylvania IRB determined there was minimal risk to participate in this study.
Arm/Group | Enhanced Electronic Platform | Electronic Platform Not Enhanced
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 0/14 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-11): https://cdn.clinicaltrials.gov/large-docs/56/NCT05207956/Prot_SAP_000.pdf